CLINICAL TRIAL: NCT00514371
Title: Phase 2/3 Randomized, Open-Label Clinical Trial of Tanespimycin (KOS-953) Plus Bortezomib Comparing Three Doses of Tanespimycin in Patients With Relapsed-Refractory Multiple Myeloma
Brief Title: A Study of Tanespimycin (KOS-953) in Patients With Relapsed-refractory Multiple Myeloma
Acronym: TIME-2
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA200-003; KAG-302
Record Dates: First submitted 2007-08-08; First posted 2007-08-09 (Estimated); Last update posted 2015-12-07 (Estimated); Status verified 2015-11

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Heat Shock Protein 90; Hsp90; KOS-953; 17-AAG; bortezomib; relapsed-refractory; tanespimycin
MeSH Terms: conditions — Multiple Myeloma | interventions — tanespimycin; Bortezomib

ARMS (3):
- tanespimycin and bortezomib (Experimental): A patient will receive a standard dose of bortezomib followed by a high dose of tanespimycin.
  Interventions: Drug: tanespimycin; Drug: Bortezomib
- bortezomib and tanespimycin (Experimental): A patient will receive a standard dose of bortezomib followed by a mid dose of tanespimycin.
  Interventions: Drug: tanespimycin; Drug: Bortezomib
- bortezomib tanespimycin (Experimental): A patient will receive a standard dose of bortezomib followed by a low dose of tanespimycin.
  Interventions: Drug: tanespimycin; Drug: Bortezomib

INTERVENTIONS:
Drug: tanespimycin — High dose
  Other Names: BMS-722782
Drug: Bortezomib — Mid dose, and low dose

SUMMARY:
This is a phase 2/3, open label trial for patients with relapsed-refractory multiple myeloma. Study agent is tanespimycin (KOS-953), at three different dose levels in combination with a fixed dose of bortezomib.

DETAILED DESCRIPTION:
Phase 2/3 combination study comparing bortezomib plus one of three doses of tanespimycin in patients with relapsed-refractory multiple myeloma after failure of at least three prior anti-cancer therapy regimens. Prior therapy must include bortezomib and lenalidomide. Primary objective is to assess the dose-response relationship of objective response rate (ORR) using EBMT/IBMTR criteria of any three dose levels of tanespimycin (KOS-953) in combination with bortezomib after four treatment cycles.

ELIGIBILITY:
Inclusion Criteria:

* Good performance status
* Histologic evidence of multiple myeloma
* Have had at least three prior treatment regimens for multiple myeloma that included both bortezomib and lenalidomide
* No prior treatment with a heat shock 90 inhibitor or an investigational proteasome inhibitor
* No known infections of HAV, HBV, HCV, or HIV
* No chemotherapy, radiation therapy, or immune therapy for three weeks prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2007-08; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate | approximately 3 months

SECONDARY OUTCOMES:
Response rate between treatment arms and time-to-event endpoints. | Up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (10):
- United States (10):
  - Local Institution, Berkeley, California
  - Local Institution, San Francisco, California
  - Local Institution, Augusta, Georgia
  - Local Institution, Baltimore, Maryland
  - Local Institution, Boston, Massachusetts
  - Local Institution, Omaha, Nebraska
  - Local Institution, New York, New York
  - Local Institution, Winston-Salem, North Carolina
  - Local Institution, Pittsburgh, Pennsylvania
  - Local Institution, Columbia, South Carolina

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx